CLINICAL TRIAL: NCT01466296
Title: Improving Treatment of People With Movement Disorders in the Middle East
Brief Title: The Middle East "Stepping Forward" Project (MESF)
Acronym: MESF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Fany Tusia, Primary Investigator: Professor Eli Lahat, Assaf-Harofeh Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HT 5283 152/09; Yad Hanadiv 5106 (Other Grant/Funding Number: Yad Hanadiv Foundation; CPIRF)
Record Dates: First submitted 2011-09-05; First posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Cerebral Palsy; Poststroke/CVA Paresis
Keywords: CERBRAL PALSY; Poststroke/CVA Paresis; REHABILITATION; WALKING; PERUTURBATION
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Re-Step (Experimental): Mechatronic shoe with a sole made to change slopes in the swing phase of walking.
  This unpredictable change will introduce a situation of necessary adaptation to keep balance
  Interventions: Device: Chaotic Perturbation
- Dummy shoes (Experimental): The shoes are in the same shape and weight of the Re-Step without the perturbations.
  Interventions: Device: Dummy not active shoes
- treadmill (Active Comparator): A treadmill with safety adaptation and all the usual characteristics of speed and slopes of fitness treadmills.
  Interventions: Device: Treadmill training

INTERVENTIONS:
Device: Chaotic Perturbation — Each subject will undergo 36 intervention sessions, 3 times per week over 12 weeks. Each session will last up to 45 minuets, depending on the subject's endurance. During each session the subject will perform basic stretching and muscle strengthening, then wear the random shoes and perform a set of exercises following specific verbal tasks, e.g., "Walk 5 strides forward," or, "Walk to the right side until I ask you to stop." During this stage of walking the device will impose perturbations in the range tolerated by the subject. The therapist will make a written report of each session.
  Other Names: Re-Step shoes
  Arms: Re-Step
Device: Dummy not active shoes — Each subject will undergo 36 intervention sessions, 3 times per week over 12 weeks. Each session will last up to 45 minuets, depending on the subject's endurance. During each session the subject will perform basic stretching and muscle strengthening, then wear the dummy shoes and perform a set of exercises following specific verbal tasks, e.g., "Walk 5 strides forward," or, "Walk to the right side until I ask you to stop." During this stage of walking the device will not impose perturbations. The therapist will make a written report of each session.
  Other Names: Dummy Shoes
  Arms: Dummy shoes
Device: Treadmill training — Each subject will undergo 36 intervention sessions, 3 times per week over 12 weeks. Each session will last up to 45 minuets, depending on the subject's endurance. During each session the subject will exercise basic stretching and muscle strengthening, then walk on the treadmill. A physiotherapist according the subject's rate of improvement will determine the increase in treadmill velocity and slope. The therapist will make a written report after each session.
  Other Names: Treadmill
  Arms: treadmill

SUMMARY:
The overall objective is to improve the functional status of Middle East adolescents with disabilities due to cerebral palsy (CP) and disabilities in adults due to cerebro-vascular stroke (Hemiplegia) by a collaborative Jordanian-Israeli-Palestinian-Moroccan applied research project.

DETAILED DESCRIPTION:
Specific objectives are:

To compare the efficacy of two rehabilitation technologies to facilitate neural reorganization, transfer and retention of treatments results to improve walking in real life situations The investigators suggest a new approach of treatment intervention that will induce unexpected changes of underfoot slopes during walking and will force the central nervous system (CNS) to react and solve problems.

The investigators also propose that the new approach will have a significantly superior motor function improvement that will be transferred to real environmental settings and be retained for long periods of time.

Research methods and materials

Subjects:

A total of 166 subjects will be studied in two groups of handicapped persons:

1. 83 Teenagers with cerebral palsy: the CP group
2. 83 Subjects with chronic hemiparesis: the HP group

Each group will be sub-divided into three secondary groups, having similar age distributions and level of motor function for the two different therapy approaches:

* 21 Treadmill exercise training
* 21 Training by randomized perturbations wearing the Random Shoe system
* 21 Training with dummy shoes without perturbations

The time flow protocol:

Recruiting subjects according to inclusion/exclusion criteria

The subjects will be tested with the following measures (see arms)at

* T0 before starting the interventions to form a base line
* T1 after 12 weeks of intensive treatments 3 x week 45 min.
* T2 6 months after T1, after the treatment was stopped, to check retainment of results of the treatments after a period of normal daily schedule of the subject

The treatments will start in a week from T0 The T1 will be performed in a week after the treatment was completed The T2 will be performed 6 months (take or leave 2 weeks) after T1, 6 months after treatment was stopped.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for CP group:

1. Diagnosis of cerebral palsy
2. Predominantly spastic type of CP with distribution of diplegia / tetraplegia
3. Age: 14 - 20 yr
4. GMFCS (gross motor function classification system) at levels II & III
5. A cognitive level sufficient to comprehend and cooperate in treatment and testing
6. No orthopedic surgery or other tone reduction intervention in last 6 months
7. Not a candidate for orthopedic surgical or other tone reduction intervention.

Exclusion criteria for CP group:

1. Candidates for orthopedic surgical or any other tone reduction procedures, e.g., botulin injections, baclofen pump interventions
2. Cannot cooperate in treatment or understand instructions
3. Uncontrolled convulsions if epileptic
4. Adolescents with progressive degenerative conditions of CNS or/and muscle-skeletal system.

Inclusion Criteria:

Inclusion criteria for HP group:

1. Stroke survivors in chronic stage (1 year or more following stroke
2. Age: 40 - 65 yr
3. Mild to moderate gait with ability to ambulate > 10m with or without assistive device
4. Cognitive level sufficient to comprehend and cooperate in tests and training
5. Mini-mental state examination (MMSE) score > 24 6: Receive medical clearance from their family physician.

Exclusion Criteria:

Exclusion criteria for HP group:

1. Dementia (Mini-Mental Score < 24)
2. Severe aphasia
3. Heart failure
4. Other medical conditions that preclude participation in low-intensity treadmill walking

Ages: 14 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
10 meter walk test (10MWT)
  10-meter walk test (Rossier & Wade, 2001) will assess normal walking speed. The participant walks a straight path distance of 10 meters at normal walking speed with time recorded. The test will be performed twice with the number of steps counted. The tester or an assistant remains near the participant to prevent a fall or injury if they appear unsteady.

SECONDARY OUTCOMES:
6 Minuets Walk Test (6MinWT)
  The 6-minute walk test (Enright, 2003) will be used to assess walking endurance. Subjects are instructed to cover as much distance as possible while walking around a marked course for 6 minutes. A member of the research staff will closely monitor the subjects.
Mechanical Efficiency
  Mechanical efficiency will be measured by the stair-climbing test (SCT) (Bar-Haim, et al. 2004; 2008). Metabolic cost is predicted from heart rate during the external work while stair-climbing and mechanical efficiency is calculated.
WHOQOL-BREF
  The WHO's Quality of Life (WHOQoL-BREF) is an international cross-culturally comparable quality of life assessment instrument. It assesses the individual's perceptions in the context of their culture and value systems, and their personal goals, standards and concerns.
Berg Balance Scale (BBS)
  The BBS is a 14-item scale that quantitatively assesses balance and risk for falls in older community-dwelling adults through direct observation of their performance.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Lahat, MD Proffesor, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Derived] Harries N, Loeppky JA, Shaheen S, Al-Jarrah M, Molteni F, Hutzler Y, Bar-Haim S; MESF Project. A stair-climbing test for measuring mechanical efficiency of ambulation in adults with chronic stroke. Disabil Rehabil. 2015;37(11):1004-8. doi: 10.3109/09638288.2014.948131. Epub 2014 Aug 12. PMID 25113573